CLINICAL TRIAL: NCT07239375
Title: Application of Intraosseous Infusion in Hematologic Critical Patients
Brief Title: Intraosseous Infusion in Hematologic Critical Patients
Status: Recruiting | Type: Observational
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanxiBethuneH4
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Intraosseous Infusions
MeSH Terms: interventions — Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: intra-osseous (IO) infusion needle/catheter — The interventional approach employed in this study is intraosseous (IO) infusion. This technique involves the percutaneous insertion of a specialized intraosseous needle or a powered driver device into the medullary cavity of a long bone (e.g., proximal tibia or humerus) to establish rapid vascular access for the administration of fluids, medications, and blood products. Its core principle leverages the bone marrow space as a "non-collapsible venous sinus," providing a rapid and effective life-saving channel for critically ill hematology patients-such as those with concomitant shock, severe hemorrhage, or multiple organ dysfunction-in whom conventional vascular access is challenging due to critical illness or underlying coagulopathies.

SUMMARY:
This single-center, prospective observational study will enroll 52 critically hematology patients aged 18-65 years including agranulocytosis, thrombocytopenia, severe anemia, advanced tumors, septic shock, sepsis DIC、 severe gastrointestinal bleeding, involvement of the central nervous system or intracranial hemorrhage, patients undergoing hematopoietic stem cell transplantation，etc. Vascular access will be established via intraosseous (IO) needle placement, primarily to evaluate first-attempt puncture success rate, therapeutic efficacy, and overall survival rate. Secondary endpoints include infusion speed, hemodynamic improvement, and procedural complications such as local infection and fat embolism. The study aims to definitively assess the efficacy and safety of IO infusion as a rapidly established, "non-collapsible" alternative vascular access route in the hematologic intensive care setting.

DETAILED DESCRIPTION:
This single-center, prospective observational study is designed to evaluate the clinical utility of intra-osseous (IO) infusion incritically hematology patients ，including:① Highly suspected or diagnosed patients with rapidly progressing highly lethal hematological diseases;② Patients with hematological disorders complicated by severe complications, including granulocyte deficiency, thrombocytopenia, severe anemia, advanced tumors, septic shock, sepsis, etc DIC、 Severe gastrointestinal bleeding, involvement of the central nervous system or intracranial hemorrhage, etc;③ Patients with hematological diseases combined with important organ dysfunction, including respiratory failure, heart failure, renal failure, liver failure, etc;④ Patients undergoing hematopoietic stem cell transplantation or those experiencing serious complications in new immunotherapy, such as hyperacute graft-versus-host disease (GVHD), grade 3-4 cytokine release syndrome (CRS) or immune effector cell associated neurotoxicity syndrome (ICANS), grade 3-4 immune checkpoint inhibitor associated interstitial lung disease, etc;⑤ Other critically patients who require life support and 24-hour monitoring.

An IO cannula will be inserted into the proximal tibia, and the following parameters will be prospectively recorded: time to vascular access, first-pass success rate, infusion flow during dwell, hemodynamic recovery, efficiency of volume resuscitation, stability of vaso-active drug delivery, and the incidence of procedure-related adverse events (local infection, fat embolism, osteomyelitis, bleeding, nerve injury). The study will explore whether IO access can serve as a reliable, rapidly established "non-collapsible" vascular route.The catheter will be removed within 24 h (maximum 96 h in exceptional cases); lidocaine step-wise analgesia will be administered according to consensus recommendations. Follow-up data will be captured in real time through an electronic case-report form (eCRF); inflammatory markers, coagulation profile, and organ-function indices will be measured by the central laboratory, while imaging specialists will assist in complication screening. The trial is intended to generate the first evidence base for IO infusion in Chinese hematology critical care and to provide feasibility and effect-size data for subsequent multicentre randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 to 65 years old. 2. Critically patients with hematologic diseases, including:① Highly suspected or diagnosed patients with rapidly progressing highly lethal hematological diseases;② Patients with hematological disorders complicated by severe complications, including agranulocytosis, thrombocytopenia, severe anemia, advanced tumors,septic shock, sepsis, DIC、 severe gastrointestinal bleeding, involvement of the central nervous system or intracranial hemorrhage, etc;③ Patients with hematological diseases combined with important organ dysfunction, including respiratory failure, heart failure, renal failure, liver failure, etc;④ Patients undergoing hematopoietic stem cell transplantation or those experiencing serious complications in new immunotherapy, such as hyperacute graft-versus-host disease (GVHD), grade 3-4 cytokine release syndrome (CRS) or immune effector cell associated neurotoxicity syndrome (ICANS), grade 3-4 immune checkpoint inhibitor associated interstitial lung disease, etc;⑤ Other critically patients who require life support and 24-hour monitoring.

Exclusion Criteria:

* 1. Fracture at the intended puncture site (due to the risk of fluid extravasation into subcutaneous tissues).

  2. Extensive soft tissue injury at the intended puncture site, resulting in insufficient anatomical landmarks for safe puncture.

  3. Local infection in the intended puncture area. 4. History of major orthopedic surgery in the intended puncture region. 5. Presence of a local prosthetic implant. 6. A site previously used for intraosseous (IO) access within the last 24 hours (to avoid re-puncture).

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study Population: Fifty-two adult patients (18-65 years) with critical hematologic disorders and poor vascular access will be enrolled. All are at imminent risk of death and include: ① rapidly progressive, highly lethal hematologic malignancies; ② severe complications such as agranulocytosis, major bleeding, DIC, CNS involvement, or sepsis; ③ concomitant respiratory, cardiac, renal, or hepatic failure; ④ life-threatening toxicities from HSCT or novel immunotherapies (hyperacute GVHD, grade 3-4 CRS/ICANS, grade 3-4 ICI-related pneumonitis); ⑤ any other critically ill patient requiring 24-h organ-supportive care.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-11-22 (Estimated); Primary Completion 2027-10-22 (Estimated); Study Completion 2027-10-23 (Estimated)

PRIMARY OUTCOMES:
First-Attempt Intraosseous Access Success Rate at 24 Hours | Assessed immediately upon IO needle placement (for success criteria) and continuously monitored for functionality for 24 hours post-placement.
  First-Attempt Intraosseous Access Success Rate at 24 Hours Defined as the proportion of patients in whom a functional intraosseous (IO) access is successfully established on the first needle insertion attempt, and which remains functional for 24 hours. Success is confirmed by: 1) Aspiration of bone marrow contents, AND 2) Free flow of saline flush without subcutaneous infiltration, AND 3) Ability to administer fluids/drugs at the desired rate.
The treatment efficacy | Assessed immediately upon IO needle placement (for success criteria) and continuously monitored for functionality for 24 hours post-placement.
  The treatment efficacy includes the recovery effect of blood routine indicators and the treatment effect of primary diseases,and overall survival rate.

SECONDARY OUTCOMES:
Overall Complication Rate Related to Intraosseous Infusion | From the time of IO access placement up to 7 days after removal, with specific assessments at 24 hours, 72 hours, and 1 month post-placement.
  Overall Complication Rate Related to Intraosseous Infusion The proportion of patients experiencing any complication attributable to the IO procedure. Complications include, but are not limited to: local pain requiring analgesia beyond the protocol-specified lidocaine, significant swelling, hematoma, subcutaneous infiltration of fluid, infection at the puncture site (assessed by redness, warmth, purulent discharge, or positive culture), osteomyelitis, compartment syndrome, limb fracture, fat embolism, or nerve injury.
Time to Achieve Hemodynamic Stability | Assessed continuously from IO access establishment until the point of hemodynamic stability is first met, up to 6 hours post-procedure.
  Time to Achieve Hemodynamic Stability ：The time interval measured from the successful establishment of IO access to the achievement of pre-defined hemodynamic stability. Stability is defined as: mean arterial pressure (MAP) ≥ 65 mmHg without increased vasopressor support, and/or heart rate (HR) decreasing to < 120 beats per minute and maintained for at least 30 minutes.
Infusion Success Rate at Target Flow Rate | Assessed during a standardized test infusion performed within 15 minutes after successful IO placement.
  The proportion of established IO accesses that are capable of delivering intravenous fluids or blood products at a clinically acceptable target flow rate (e.g., ≥ 100 mL/min for tibial site or ≥ 150 mL/min for humeral site) without failure (e.g., dislodgement, occlusion, or significant leakage).
30-day All-Cause Mortality | From the date of IO access placement up to 30 days.
  The proportion of patients who die from any cause within 30 days following the establishment of intraosseous access.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China